CLINICAL TRIAL: NCT01792102
Title: A Phase 1/2 Study of Safety, Efficacy, and Pharmacodynamics of a 60-Minute Infusion of Carfilzomib for Patients With Progressive Multiple Myeloma
Brief Title: Safety, Efficacy, and Pharmacodynamics of a 60-Minute Infusion of Carfilzomib for Progressive Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oncotherapeutics (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-CAR-585
Record Dates: First submitted 2013-01-03; First posted 2013-02-15 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Carfilzomib; Krypolis; 60 minute infusion
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib and Dexamethasone (Experimental): Phase 1: Carfilzomib will be administered at an escalating dose with dexamethasone administered at 8mg.
  Phase 2: Carfilzomib will be administered at the MTD determined in phase 1. Maintenance: Carfilzomib and dexamethasone will be administered in the same fashion as the previous treatment cycles, but only on days 1, 2, 15, and 16.
  Interventions: Drug: Carfilzomib and Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib and Dexamethasone — Phase 1: Carfilzomib will be administered at an escalating dose by cohort as 60-minute IV infusion on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle. On Cycle 1 Days 1 and 2, carfilzomib will be given at 20 mg/m^2. For all subsequent doses, carfilzomib will be administered at the dose assigned to the cohort (56, 70, or 88 mg/m^2). Dexamethasone (8 mg IV or PO) will be administered prior to carfilzomib on Days 1, 2, 8, 9, 15, and 16.
  Phase 2: Carfilzomib will be administered at the MTD determined in phase 1. Maintenance: From Cycle 9 onward, carfilzomib and dexamethasone will be administered in the same fashion as during the previous treatment cycle, but only on days 1, 2, 15, and 16.
  Other Names: Krypolis®

SUMMARY:
This is a Phase 1/2, multicenter, open label, dose-escalation, nonrandomized study to evaluate the safety, pharmacodynamics, and efficacy of a 60-minute infusion of carfilzomib for patients with progressive multiple myeloma.

DETAILED DESCRIPTION:
This is a Phase 1/2, multicenter, open label, dose-escalation, nonrandomized study to evaluate the safety, pharmacodynamics, and efficacy of a 60-minute infusion of carfilzomib for patients with progressive multiple myeloma.

The study will consist of a screening period, followed by a treatment period of up to eight 28-day treatment cycles, followed by a period of maintenance treatment. Subjects are to be treated until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. MM with relapsing or progressive disease at study entry

   a. Defined as progressive MM on patient's last treatment regimen
2. Measurable disease, as defined by one or more of the following (assessed within 14 days prior to first dose):

   1. Serum M-protein ≥ 0.5 g/dL, or
   2. Urine M-protein ≥ 200 mg/24 hours, or
   3. Only in patients who do not meet a or b, then use serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal kappa/lamda ratio
3. Age ≥ 18 years
4. Life expectancy ≥ 6 months
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Adequate hepatic function within 14 days prior to first dose, with bilirubin < 1.5 × the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 × ULN
7. LVEF ≥ 40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Multigated Acquisition Scan (MUGA) is acceptable if ECHO is not available.
8. Absolute neutrophil count (ANC) ≥ 1000/mm3 within 14 days prior to first dose. Screening ANC is to be independent of granulocyte colony stimulating factor support for ≥ 1 week and pegylated granulocyte colony stimulating factor for ≥ 2 weeks.
9. Hemoglobin ≥ 8.0 g/dL within 14 days prior to enrollment. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed.
10. Platelet count ≥ 75,000/mm3 (≥ 50,000/mm^3 if myeloma involvement in the bone marrow is > 50%) within 14 days prior to first dose. Patients must not have received platelet transfusions for at least 7 days prior to obtaining the screening platelet count
11. Calculated or measured creatinine clearance (CrCl) of ≥ 15 mL/min within 14 days prior to first dose. Calculation are based on a standard formula, such as the Cockcroft and Gault: [(140 - Age) x Mass (kg) / (72 x Creatinine mg/dL)]; multiply result by 0.85 if female
12. Written informed consent in accordance with federal, local, and institutional guidelines
13. Female patients of childbearing potential (FCBP) must have a negative serum pregnancy test within 14 days prior to first dose and agree to use an effective method of contraception during and for 3 months following last dose of drug (more frequent pregnancy tests may be conducted if required per local regulations). Postmenopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from a pregnancy test
14. Male patients must agree to use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with a FCBP

Exclusion Criteria:

1. Multiple myeloma of IgM subtype
2. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
3. Plasma cell leukemia (> 2.0 × 109/L circulating plasma cells by standard differential)
4. Waldenström's macroglobulinemia
5. Amyloidosis
6. Glucocorticoid therapy (prednisone > 30 mg/day or equivalent) within 7 days prior to first dose
7. Cytotoxic chemotherapy with approved or investigational anticancer therapeutics within 28 days prior to first dose
8. Treatment with bortezomib, thalidomide or lenalidomide within 21 days prior to first dose
9. Focal radiation therapy within 7 days prior to first dose. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to enrollment (i.e., prior radiation must have been to < 30% of the bone marrow)
10. Immunotherapy within 21 days prior to first dose
11. Major surgery within 21 days prior to first dose
12. Active congestive heart failure (New York Heart Association [NYHA] Classes III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 6 months prior to first dose.
13. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at HBV), or antifungal agents within 14 days prior to first dose
14. Known human immunodeficiency virus (HIV) seropositivity
15. Known hepatitis B or C virus infection (except for patients with HBV receiving and responding to HBV antiviral therapy: these patients are allowed)
16. Patients with known cirrhosis
17. Second malignancy within the past 3 years, except:

    1. Adequately treated basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
    3. Prostate cancer < Gleason score 6 with stable prostate-specific antigen (PSA) over 12 months
    4. Breast carcinoma in situ with full surgical resection
    5. Treated medullary or papillary thyroid cancer
    6. Patients with myelodysplastic syndrome
18. Significant neuropathy (Grades 3 to 4) within 14 days prior to first dose
19. Peripheral neuropathy with pain ≥ G2 within 14 days prior to first dose
20. Female patients who are pregnant or lactating
21. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
22. Prior carfilzomib treatment
23. Prior participation in any Onyx-sponsored phase 3 trial
24. Patients with contraindication to dexamethasone
25. Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
26. Ongoing graft-versus-host disease
27. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrollment
28. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment
29. Any other clinically significant medical disease or psychiatric condition that, in the Investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2013-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Establish maximum tolerated dose (MTD) | monthly, up to 24 months
  Maximum tolerated dose will be established by the number of dose limiting toxicities and the overall safety and tolerability of the study drug.
  Safety and tolerability will be determined by the following:
  1. incidence and frequency of adverse events throughout the study
  2. clinical laboratory test results at study visits
  3. vital signs measurements at each study visits
  4. medical history and physical examination findings
  5. ECOG performance status at study visits
  6. concomitant medication usage throughout the study

SECONDARY OUTCOMES:
Establish efficacy as assessed by the overall response rate | monthly, up to 24 months
  Response rate will be determined by the following:
  1. SPEP, UPEP, and quantification of immunoglobulins and immunofixation
  2. bone marrow aspirates and biopsies to confirm CR
  3. roentgenographic skeletal survey
  Response rate will be assessed by the following:
  1. Clinical benefit response rate
  2. Progression-free survival
  3. Time to progression
  4. Duration of response
  5. Overall survival
  6. Pharmacodynamics

OTHER OUTCOMES:
Relationship of 60-minute infusion of carflizomib with pharmacodynamic markers | weekly for 2 months

CONTACTS AND LOCATIONS:
Overall Officials: James Berenson, M.D., Principal Investigator — James Berenson Inc.; Joshua Richter, M.D, Principal Investigator — John Theurer Cancer Center at Hackensack University Medical Center
Locations (2):
- United States (2):
  - James R. Berenson M.D. Inc., West Hollywood, California
  - John Theuer Cancer Center Hackensack University Medical Center, Hackensack, New Jersey